CLINICAL TRIAL: NCT05109767
Title: The Effect of Virtual Reality Glass and Smartphone Game Application on Preoperative Anxiety in 7-13 Years Children
Brief Title: The Effect of Virtual Reality Glass and Smartphone Game Application on Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nuray Caner, Lecturer, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/103
Record Dates: First submitted 2021-10-08; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality glass game application (Experimental)
  Interventions: Device: Virtual reality
- Smartphone game application (Active Comparator)
  Interventions: Device: Smartphone
- Control group (No Intervention)

INTERVENTIONS:
Device: Virtual reality — The Virtual Reality Glass game application reduces anxiety by distracting attention..The virtual reality glass game was played to intervention group for 15 minutes before surgery.
  Arms: Virtual reality glass game application
Device: Smartphone — The Smartphone game application reduces anxiety by distracting attention. Smartphone game was played to intervention group for 15 minutes before surgery.
  Arms: Smartphone game application

SUMMARY:
This study was conducted to evaluate the effects of virtual reality glasses and smartphone game applications on preoperative anxiety in children who have day surgery. The study comprised of 60 children (20 children in a virtual reality glass game application group, 20 children in a smartphone game application group, and 20 children in a control group). The approval of the ethics committee, permissions from the institutions, and informed voluntary approval of the children's were obtained to conduct the research. The data of the research were collected through the Children's Perioperative Multidimensional Anxiety Scale (CPMAS), physiological parameters of children were measured before, after and 90 minutes after the operation, and salivary cortisol sample taken before surgery in all of groups. Children in smartphone game application groups played a game for 15 minutes on a smartphone before the surgical operation, and standard care was given to children. Children in virtual reality game application groups played a game for 15 minutes on virtual reality glasses before the surgical operation, and standard care was given to children. Before the surgical operation, standard care was given to children in control groups. The value of p<0.05 was accepted statistically significant in the data analyses.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted to evaluate the effects of virtual reality glasses and smartphone game applications on preoperative anxiety in children who have day surgery. The study was performed between the ages of 7-13 years children at a tertiary hospital. Age, gender, surgery type, previous hospitalization experience and having chronic disease criteria of the children in control group (n=20), smartphone game application (n=20) and virtual reality glass game application (n=20) groups. Data were collected with Descriptive Characteristics Form for Children and Families, Children's Perioperative Multidimensional Anxiety Scale (CPMAS). Before the surgical operation, the game with a smartphone and virtual reality glass was played to the intervention groups for 15 minutes. Physiological parameters of children were measured before, after and 90 minutes after the operation. In addition, CPMAS was applied to children in preoperative assessment (Time 1), on the day of the operation (Time 2) and one month postoperatively (Time 3). Data were analyzed with post-power analysis, descriptive statistics, Kruskal-Wallis and Friedman Tests. The value of p<0.05 was accepted statistically significant in the data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Between 7 and 13 years of age
* Patients scheduled for day surgery
* Not having vision, hearing or speech problems
* Understands the Turkish language
* Not having a mental or neurological disability
* Not having a history of convulsions

Exclusion Criteria:

* Does not understand the Turkish language
* the child is under 7 years old or 13 years older
* having vision, hearing or speech problems
* having a mental or neurological disability
* having a history of convulsions

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Children's Perioperative Multidimensional Anxiety Scale (CPMAS) Mean Score | An average of 45 days: In preoperative assessment (Time 1), on the day of the operation (Time 2) and one month postoperatively (Time 3).
  According to the CPMAS, a score between 0-500 is obtained from the scale. A high score from the scale indicates a high level of perioperative anxiety. Change= in preoperative assessment (Time 1), on the day of the operation (Time 2) and one month postoperatively (Time 3).

SECONDARY OUTCOMES:
Physiological parameters | One day: One day: Half an hour before and, 45 minutes before the operation and 90 minutes after the operation.
  Heart Rate, Change= Half an hour before and, 45 minutes before the operation and 90 minutes after the operation.
Physiological parameters | One day: Half an hour before and, 45 minutes before the operation and 90 minutes after the operation.
  Oxygen saturation, Change= Half an hour before and, 45 minutes before the operation and 90 minutes after the operation.
Physiological parameters | One day: One day: Half an hour before and, 45 minutes before the operation and 90 minutes after the operation.
  Blood pressure, Change= Half an hour before and, 45 minutes before the operation and 90 minutes after the operation.

OTHER OUTCOMES:
Salivary cortisol | One day: Half an hour before the operation
  Serum biochemical parameters.The high level of salivary cortisol is interpreted as an increase in cortisol secretion.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Caner, Dr, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No